CLINICAL TRIAL: NCT05683730
Title: Intermittent Caloric Restriction in Patients With Mild to Moderate Crohn's Disease: A Randomized, Open-label, Controlled Trial
Brief Title: Intermittent Caloric Restriction in Patients With Mild to Moderate Crohn's Disease
Acronym: TONIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, CARON Bénédicte, Doctor, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-A02169-34
Record Dates: First submitted 2022-12-20; First posted 2023-01-13 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Crohn's Disease
Keywords: intermittent caloric restriction; Crohn's disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent caloric restriction (Experimental): Intermittent caloric restriction during 16 weeks.
  Interventions: Other: Intermittent caloric restriction
- Routine practice (No Intervention): Routine practice

INTERVENTIONS:
Other: Intermittent caloric restriction — Intermittente caloric restriction:
  1. st month: restriction of 50% of the caloric intake previously determined by the dietician 1 day per week
  2. nd month: restriction of 50% of the caloric intake 2 days per week
  3. rd month: restriction of 60% of the caloric intake 2 days per week
  4. th month: restriction of 75% of the caloric intake 2 days per week
  Arms: Intermittent caloric restriction

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory disease of the gastrointestinal (GI) tract. CD is a common inflammatory bowel disease (IBD), frequent (150,000 patients in France and 1.5 million in Europe), disabling and incurable. The environmental factors, and in particular diet, play a major role in the pathogenesis of CD. The prevalence of CD is steadily increasing in highly industrialized countries, where the Western diet rich in saturated fats and refined sugars, is blamed for this to explain this true pandemic. On the other hand, enteral nutrition, exclusive or partial, is known to be effective in the initial treatment of CD, especially in pediatrics.

There are a number of evidence in favor of a nutritional management nutritional management of caloric restriction during inflammatory diseases such as psoriasis and rheumatoid arthritis,whose physiopathology is similar to that of IBD.

To date, and despite patient concern, there is no consensus nutritional in the management of CD to influence the natural course of the disease.

The investigators have decided to initiate a clinical study to evaluate for the first time the efficacy, acceptability and safety of intermittent caloric restriction in patients with CD.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 65 years old
* Established diagnosis of Crohn's disease with a minimum disease duration of 3 months
* Patient with mild to moderate Crohn's disease defined by a fecal calprotectin ≥ 250 μg/g and a CDAI score between 150 to 300
* Medical treatment of Crohn's disease stable for at least 3 months
* Patient compliant with an intermittent caloric restriction during 16 weeks
* Person affiliated to or beneficiary of a social security plan
* Person informed about study organization and having signed the informed consent

Exclusion Criteria:

* Patient with a BMI < 18.5kg/m2
* Patient having a weight loss of 5% the first month and 10% during the first 6 months
* Patient with active ano-perineal lesions
* Patient with an ostomy
* Patient with eating disorders (anorexia, bulimia)
* Person referred in articles L.1121-5, L. 1121-7 and L.1121-8 of the Public Health Code:

  * Pregnant, parturient or breastfeeding woman
  * Minor person (non-emancipated)
  * Adult person under legal protection (any form of public guardianship)
  * Adult person incapable of giving consent and not under legal protection
* Person deprived of liberty for judicial or administrative decision, person under psychiatric care as referred in articles L. 3212-1 and L. 3213-1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Intestinal inflammation | week 16
  Evaluate the effectiveness of personalized nutritional management of intermittent caloric restriction during 16 weeks on the level of intestinal inflammation (induction of of a biological response) in patients with mild to moderate CD mild to moderate. The effectiveness will be evaluated in each group by a biological response change, that is to say a decrease at least 50% of calprotectin fecal level.

SECONDARY OUTCOMES:
Induction of a clinical response | week 16
  Evaluate the impact of personalized nutritional management of intermittent caloric restriction during 16 weeks on Crohn's Disease Activity Index (CDAI) that is to say change by al least 100 points.
  The following cut-offs correlate with level of disease activity:
  Non-active disease: CDAI < 150 Mild disease activity: CDAI >= 150 and <220 Moderate disease activity: CDAI >= 220 and <450 Severe disease activity: CDAI > 450
Induction of a clinical remission | week 16
  Evaluate the impact of personalized nutritional management of intermittent caloric restriction during 16 weeks on clinical remission, that is to say Crohn's Disease Activity Index (CDAI) < 150
  The following cut-offs correlate with level of disease activity:
  Non-active disease: CDAI < 150 Mild disease activity: CDAI >= 150 and <220 Moderate disease activity: CDAI >= 220 and <450 Severe disease activity: CDAI > 450
Induction of a biological remission | week 16
  Evaluate the impact of personalized nutritional management of intermittent caloric restriction during 16 weeks on biological remission that is to say fecal calprotection < 250 µg/g
Induction of a radiological response | week 16
  Evaluate the impact of personalized nutritional management of intermittent caloric restriction during 16 weeks on radiological response that is to say change of 50% of Nancy score measured by magnetic resonance imaging (MRI)
  Total MRI score: 0 at 36
Improving quality of life | week 16
  Evaluated by short-Inflammatory Bowel Disease Questionnaire (short-IBDQ)
  short-IBDQ is a 10-items measure that assesses self-reported quality of life. Total score ranges from 10 to 70. Higher the score is better life quality is.
Improving work productivity | week 16
  Evaluated by Work Productivity and Activity Impairment Questionnaire (WPAI)
  WPAI questions measure the effect of patients health problems (any physical or emotional problem or symptom) on their ability to work and perform regular activites.
Improving fatigue | week 16
  Evaluated by Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
  FACIT-F is a 40-items measure that assesses self-reported fatigue and its impact upon daily activities and function.
Improving functional disability | week 16
  Evaluated by Inflammatory Bowel Disease - Disability Index (IBD-DI)
  IBD-DI is a 14-items measure that assesses self-reported disability. It ranges from 0-100: 0-20 (no disability), 20-35 (mild disability), 35-50 (moderate disability) and 50-100 (severe disability)
Improving anxiety disorder | week 16
  Evaluated by Generalized Anxiety Disorder (GAD-7)
  The following cut-offs correlate with level of anxiety severity:
  Score 0-4: Minimal Anxiety Score 5-9: Mild Anxiety Score 10-14: Moderate Anxiety Score greater than 15: Severe Anxiety
Evaluate the safety of intermittent caloric restriction in patients with mild to moderate with mild to moderate CD. | weeks 4;8;12 and 16
  Percentage of adverse event related to intermittent caloric restriction (fatigue; nausea; headache, dizziness, hypotension, irritability, capacity reduced to concentrating, undernutrition/sarcopenia)
Evaluate compliance of intermittent caloric restriction during 16 weeks in patients with with mild to moderate CD. | week 16
  Percentage of patient compliance measured by for example a intermittent caloric restriction during at least 21 days on the 16 weeks of the study
Determine the level of patient satisfaction with intermittent caloric restriction | week 16
  Evaluated by Likert scale at 4 items ad-hoc
  4 point likert scale for the frequency; assign each response a point value from 1 to 4.
Estimate, in the experimental arm, the prevalence of compensatory hyperphagia after intermittent caloric restriction | 48 hours after intermittent caloric restriction
  Percentage of patients having a compensatory hyperphagia after 2 days of intermittent caloric restriction.

CONTACTS AND LOCATIONS:
Overall Officials: CARON Bénédicte, MD, Principal Investigator — CHRU of Nancy, Hepatogastroenterology Department
Locations (1):
- CHRU of Nancy, Vandœuvre-lès-Nancy, CHRU de Nancy, France

REFERENCES:
- [Background] Yanai H, Levine A, Hirsch A, Boneh RS, Kopylov U, Eran HB, Cohen NA, Ron Y, Goren I, Leibovitzh H, Wardi J, Zittan E, Ziv-Baran T, Abramas L, Fliss-Isakov N, Raykhel B, Gik TP, Dotan I, Maharshak N. The Crohn's disease exclusion diet for induction and maintenance of remission in adults with mild-to-moderate Crohn's disease (CDED-AD): an open-label, pilot, randomised trial. Lancet Gastroenterol Hepatol. 2022 Jan;7(1):49-59. doi: 10.1016/S2468-1253(21)00299-5. Epub 2021 Nov 2. PMID 34739863
- [Background] Jiang Y, Jarr K, Layton C, Gardner CD, Ashouri JF, Abreu MT, Sinha SR. Therapeutic Implications of Diet in Inflammatory Bowel Disease and Related Immune-Mediated Inflammatory Diseases. Nutrients. 2021 Mar 10;13(3):890. doi: 10.3390/nu13030890. PMID 33801883